CLINICAL TRIAL: NCT05136846
Title: A Phase I Trial Targeting Mitochondrial Metabolism With Papaverine in Combination With Chemoradiation for Stage II-III Non-Small Cell Lung Cancer
Brief Title: Papaverine in Combination With Chemoradiation for the Treatment of Stage II-III Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeremy Brownstein, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20327; NCI-2021-07691 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA262388 (NIH)
Record Dates: First submitted 2021-08-17; First posted 2021-11-29 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Lung Non-Small Cell Carcinoma; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Unresectable Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; durvalumab; Immunoglobulin G; Disulfides; Paclitaxel; Taxes; Papaverine; Radiotherapy; Radiation; Pemetrexed; Radiation Dose Hypofractionation; Magnetic Resonance Spectroscopy; X-Rays; Contrast Media; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (papaverine, RT, paclitaxel, carboplatin) (Experimental): Patients receive PPV IV or SC over 30 minutes and patients receiving chemoradiation undergo 5 fractions of RT per week for 6 weeks or 5 fractions of hypofractionated RT per week for 3 weeks without chemotherapy. Patients undergoing chemoradiation receive paclitaxel IV and carboplatin IV QW over 1-6 weeks or pemetrexed IV followed by carboplatin IV every 3 weeks during radiation in the absence of disease progression or unacceptable toxicity. Patients with PD-L1 positive disease may also receive durvalumab after completing CRT as considered clinically appropriate by the treating medical oncologist. Patients also undergo PET/CT or CT and brain MRI during screening, and blood sample collection, MRI and CT scans throughout the trial.
  Interventions: Drug: Carboplatin; Biological: Durvalumab; Drug: Paclitaxel; Drug: Papaverine; Radiation: Radiation Therapy; Drug: Pemetrexed; Radiation: Hypofractionated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging of the Brain with and without Contrast; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Papaverine — Given IV or SC
  Other Names: Cerebid; Cerespan; Pavabid; Pavacap; Pavatym; Robaxapap
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated RT
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging; PET; Pet Scan; Positron emission tomography (procedure); positron emission tomography scan; Positron-Emission Tomography; PT
Procedure: Computed Tomography — Undergo PET/CT or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT SCAN; tomography
Procedure: Magnetic Resonance Imaging of the Brain with and without Contrast — Undergo brain MRI
  Other Names: Brain Magnetic Resonance Imaging with and without Contrast; Brain MRI; Brain MRI with and without Contrast; Head MRI with and without Contrast
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase I trial finds out the best dose, possible benefits and/or side effects of papaverine when given together with chemoradiation intreating patients with stage II-III non-small cell lung cancer. Papaverine targets mitochondrial metabolism to decrease the cancer growth process. Giving papaverine with chemoradiation may work best to treat patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximally tolerated dose of papaverine (PPV) in combination with chemoradiation (CRT)/radiation therapy (RT) in patients with unresectable locally advanced (LA) non-small cell lung cancer (NSCLC) or oligometastatic NSCLC.

SECONDARY OBJECTIVES:

I. To estimate the rates of primary tumor control, local control, time to local-regional progression, disease-free survival (DFS), and overall survival (OS). II. To assess whether blood oxygen level determination (BOLD) functional magnetic resonance imaging (MRI) studies can predict which patients may respond best to PPV + CRT/RT, and detect changes in oxygenation before and after PPV administration.

III. To assess whether blood-based and tissue-based biomarkers can predict which patients may respond best to PPV + CRT.

OUTLINE: This is a dose-escalation study of PPV.

Patients receive PPV intravenously (IV) or subcutaneously (SC) over 30 minutes and patients receiving chemoradiation undergo 5 fractions of radiation therapy (RT) per week for 6 weeks or 5 fractions of hypofractionated RT per week for 3 weeks without chemotherapy. Patients undergoing chemoradiation receive paclitaxel IV and carboplatin IV once weekly (QW) over 1-6 weeks or pemetrexed IV followed by carboplatin IV every 3 weeks during radiation in the absence of disease progression or unacceptable toxicity. Patients with PD-L1 positive disease may also receive durvalumab after completing CRT as considered clinically appropriate by the treating medical oncologist. Patients also undergo positron emission tomography/computed tomography (PET/CT) or CT and brain magnetic resonance imaging (MRI) during screening, and blood sample collection, MRI and CT scans throughout the trial.

After completion of the study treatment, patients are followed for 2 years at 1, 3, 6, 9, 12, 16, 20, and 24 months, then periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0) =< grade 1 (except alopecia) at the time of enrollment
* Absolute neutrophil count >=1.5 x 10^9/L
* Hemoglobin >= 9 g/dL
* Platelets >= 100 x 10^9/L
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine < 1.5 mg/dL or calculated creatinine clearance* >= 50 mL/min or 24-hour urine creatinine clearance >= 50 mL/min

  * Calculated by the Cockcroft-Gault formula •>= 18 years old
* Non-small cell lung cancer (NSCLC), histologically and/or cytologically proven
* Clinical American Joint Committee on Cancer (AJCC) stage II-III NSCLC (T1-4N0-3M0) and select patients with stage IV oligometastatic disease.

  * For patients with oligometastatic disease (up to 5 total sites of disease) for whom definitive CRT or RT to the primary and regional lymph nodes is recommended by the multidisciplinary team, each individual metastatic tumor would be considered an additional site of disease with the exception of brain metastases. Up to 10 brain metastases would be considered as 1 site.
  * Patients with oligometastatic disease will be allowed to receive adjuvant systemic therapy at the discretion of the medical oncologist and additional local therapy to metastatic sites at the discretion of the multidisciplinary team
* Patients must be considered unresectable or medically-inoperable if stage II-III NSCLC

  * Patients with a local or regional recurrence following surgical resection for whom definitive CRT or RT to disease in the chest is recommended by the multidisciplinary team will be considered eligible
* Patients must have fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)-computed tomography (CT) scan (or CT chest/abdomen/pelvis with IV contrast), and magnetic resonance imaging (MRI) brain with IV contrast (preferred) or CT scan of the brain with contrast. Non-contrast MRI scans of the chest/abdomen/pelvis or brain are permitted for workup if patient has allergy to CT contrast or renal insufficiency
* Patients must have vital signs, history/physical examination, laboratory studies (complete blood count [CBCP] with differential, chemistries including liver function tests, creatinine clearance (CrCl) assessment; pregnancy test if needed within 14 days of registration)
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* No history of complete atrioventricular block, hepatic dysfunction (e.g. cirrhosis), glaucoma, or priapism
* Patients must be a minimum of 3 weeks from thoracotomy (if performed) and well-healed before starting treatment
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test within 14 days of registration. Urine human chorionic gonadotropin (HCG) is an acceptable pregnancy assessment
* Nursing women may participate only if nursing is discontinued, due to the possibility of harm to nursing infants from the treatment regimen
* Women/men of reproductive potential must be counselled on contraception/ abstinence while receiving the study treatment

  * Women of childbearing potential are required to use an effective method of contraception from the time of negative serum pregnancy test, throughout the study duration, and until 4 years after the last dose of radiation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
  * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 6 months after completion of study drug administration
* For patients planning to undergo CRT, patient is suitable to receive standard chemotherapy per treating medical oncologist with radiation during study treatment

INCLUSION CRITERIA FOR MRI IMAGING SUB-STUDY:

•Patients must consent to participate in the main part of this study and be enrolled into the expansion cohort, or consent to participate in the main part of this study and also consent to participate in the optional MRI Imaging study

Exclusion Criteria:

* Patients with history of pneumonectomy
* History of active connective tissue disease (scleroderma) or idiopathic pulmonary fibrosis
* History of previous radiation therapy which would result in overlapping radiation fields
* Subjects who are breast-feeding and plan to continue breast-feeding during therapy, or have a positive pregnancy test will be excluded from the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Hepatic insufficiency resulting in jaundice, or not meeting laboratory values above (albumin, total bilirubin, AST/ALT)
* Patients enrolled into the expansion cohort must be able to complete the MRI Sub-study, or at a minimum attempt the first scan of the MRI Sub-study
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the treating physicians. This could include severe, active co-morbidities such as:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acquired immune deficiency syndrome (AIDS) based upon the current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration
* Patients who are presently receiving nitrates or nitroglycerin, or have received these medications within 30 days of day 1 of protocol treatment
* Patients who are currently taking Sildenafil should agree to discontinue use for 2 days prior to initiation of papaverine, during the duration of study, and for 2 days after last dose of papaverine

EXCLUSION CRITERIA FOR MRI IMAGING SUB-STUDY:

* Any medical contraindication to MR imaging (e.g. pacemakers, metallic implants, aneurysm clips, pregnancy, nursing mothers, weight greater than 350 pounds)
* Severe anxiety/claustrophobia related to MR imaging despite medications to relieve anxiety/claustrophobia
* Patients who use supplemental oxygen and are not able to stop their oxygen for up to a few hours at a time, or who use oxygen because they have breathing when they are laying down

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximally tolerated dose (MTD) of papaverine (PPV) in combination with chemoradiation treatment (CRT) or definitive hypofractionated radiation therapy | 6 weeks
  Will employ the Time-to-event Bayesian optimal interval design to find the MTD. Treatment-related toxicity will be assessed based on Common Terminology Criteria for Adverse Events version 5.0 criteria.

SECONDARY OUTCOMES:
Primary tumor control rate | At 12 and 24 months post-treatment
  Defined as the absence of primary tumor failure. Will be calculated and 95% exact binomial confidence interval will be provided.
Local control rate | At 12 and 24 months post-treatment
  Defined as the absence of local failure, which is a combination of primary tumor and involved lobe failure. Will be calculated and 95% exact binomial confidence interval will be provided.
Time to local-regional progression | From entry on the study until the time of documented local-regional recurrence or death, assessed at 12 and 24 months post-treatment
  Will be summarized using Kaplan-Meier method.
Disease-free survival | From entry on the study until the time of any documented disease recurrence or death, assessed at 12 and 24 months post-treatment
  Will be summarized using Kaplan-Meier method.
Distant-metastasis-free survival | At 12 and 24 months post-treatment
  Will be summarized using Kaplan-Meier method.
Overall survival | From study entry until the time of death from any cause, assessed at 12 and 24 months post-treatment
  Will be summarized using Kaplan-Meier method.
Changes in magnetic resonance imaging (MRI) blood oxygen level dependent (BOLD) response on MRI | Baseline up to 24 months
  Images pre and post PPV will be analyzed for stability of baseline and treatment signals. Percent BOLD change will be determined for maximal and overall signal changes. Comparisons between the distributions of pre and post PPV will be valuated using Earth Mover's Distance.
Changes in blood-based biomarkers related to predict patients response to PPV + CRT | Baseline up to 24 months
  Will acquire measurements of circulating serum microRNAs that can indicate tumor hypoxia or response to therapeutic intervention, and alterations in immune cell subsets that are suggestive of immune system activation or suppression with the experimental therapy
Changes in tissue-based biomarkers related to predict patients response to PPV + CRT | Baseline up to 24 months
  When biopsy tissue is available, will acquire gene expression profiles by Affymetrix gene chip for indications of tumor hypoxia or response to therapeutic intervention, and correlating tumor mutations in genes involved in the anti-oxidant response pathway with outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremey Brownstein, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu